CLINICAL TRIAL: NCT05610085
Title: A Phase IIb Dose Escalation Study of Levetiracetam for the Treatment of Neonatal Seizures
Brief Title: A Dose Escalation Study of Levetiracetam in the Treatment of Neonatal Seizures
Acronym: NEOLEV3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Minnesota (Other); Rady Children's Hospital, San Diego (Other); Auckland City Hospital (Other Government); University of Auckland, New Zealand (Other); Middlemore Hospital, New Zealand (Other)
Responsible Party: Principal Investigator, Richard H. Haas, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-6335
Record Dates: First submitted 2022-10-27; First posted 2022-11-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Neonatal Seizure; Neonatal Encephalopathy; Hypoxic-Ischemic Encephalopathy; Seizure Newborn
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Levetiracetam; Phenobarbital

STUDY DESIGN:
Intervention Model Description: If seizures persist or recur after 60 mg/kg LEV patients will be randomized to receive either dose escalation of levetiracetam or phenobarbital. Randomization will occur in a 3:1 ratio LEv: PHB stratified by site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation with LEV (Experimental): Additional LEV at a higher dose (30 mg/kg, 60 mg/kg, or 90 mg/kg depending on the stage of the study).
  Interventions: Drug: Levetiracetam Injection
- Standard of care Phenobarbital (Active Comparator): Treatment with Phenobarbital 20mg/kg IV and if needed a further 20mg/kg totalling 40mg/kg
  Interventions: Drug: Phenobarbital Sodium Injection

INTERVENTIONS:
Drug: Levetiracetam Injection — Neonates will be treated with intravenous levetiracetam 60mg/kg for first line management of seizures, and if seizures persist will be randomized to receive higher dose Levetiracetam or standard of care phenobarbital
  Arms: Dose escalation with LEV
Drug: Phenobarbital Sodium Injection — Standard of care for neonatal seizures
  Arms: Standard of care Phenobarbital

SUMMARY:
The main purpose of this study is to determine the maximum safe tolerated dose of LEV in the treatment of neonatal seizures. Our hypothesis is that optimal dosing of Levetiracetam (LEV) to treat neonatal seizures is significantly greater than 60mg/kg. This study will be an open label dose-escalation, preliminary safety and efficacy study. There will be a randomized control treatment component. Infants recognized as having neonatal seizures or as being at risk of developing seizures will be recruited and started on continuous video EEG monitoring (CEEG). Eligibility will be confirmed and consent will be obtained. In the first 2 phases of the study, neurologists will identify neonates with mild-moderate seizure burden (less than 8 minutes cumulative seizure activity per hour), appropriate for study with LEV, and exclude patients with higher seizure burden where treatment with PHB is more appropriate. Phase 3 of the dose escalation will only proceed if additional efficacy of LEV has been demonstrated in phases 1 and 2. In Phase 3 we will recruit neonates with seizures of greater severity up to 30 minute seizure burden/hour. This will make the final results of study more generalizable.

If seizures are confirmed, enrolled subjects will receive 60mg/kg of LEV. Subjects whose seizures persist or recur 15 minutes after the first infusion is complete, subjects will then be randomized in the dose escalation study. Patients in the dose escalation study will be randomly assigned to receive either higher dose LEV or treatment with the control drug PHB in a 3:1 allocation ratio, stratified by site.

Funding Source- FDA OOPD

DETAILED DESCRIPTION:
Aims/Hypotheses:

Primary Aim: To determine the recommended maximal safe dose of LEV in the setting of neonatal seizures of mild to moderate severity.

If 60mg/kg LEV does not control seizures, subjects will be randomised to receive either additional LEV or PHB. LEV dose will be escalated in 30mg/kg increments to a maximal dose of 150mg/kg total loading dose. We will use a continual reassessment method to determine the maximal safe and tolerated dose.

Secondary/exploratory aims:

* To study the pharmacokinetics of high dose LEV in neonates with seizures of mild to moderate severity.
* To estimate the additional efficacy of higher doses of LEV in neonates with seizures of mild to moderate severity.
* To improve technologies for the prompt detection of neonatal seizures: We will assess the latest version of Persyst's neonatal seizure detector.

Research Design

This is a Phase IIb, open label dose-escalation, preliminary safety and efficacy study. An active drug treatment control arm (PHB group) is included in the study design. This study is not designed or powered to compare high dose LEV and PHB groups, however, the randomized control group will help with interpretation of adverse events and seizure cessation efficacy seen in the high dose escalation group. This is particularly important because of the high rates of morbidity in neonates with seizures.

24-hour seizure control endpoint: cEEG reviewed by a neurophysiologist will be used for assessing 24-hour seizure control. Treatment will be considered effective in achieving 24-hour seizure control if there is a seizure burden less than 30 seconds in the 24 hours following the dose. Change in seizure burden in 2-hour post treatment period will also be assessed.

Intervention If seizure activity occurs participants will be enrolled and will receive 60mg/kg LEV.

If seizures continue babies will then be randomised to receive either:

* Additional LEV at a higher dose (30 mg/kg, 60 mg/kg, or 90 mg/kg depending on the stage of the study), OR
* PHB at 20-40 mg/kg. Maintenance treatment will continue for 5 days, either IV or orally if baby is tolerating feeds.

LEV discontinuation or addition of PHB: there are multiple criteria for transition to, or addition of, PHB treatment if required for seizure control.

ELIGIBILITY:
Inclusion Criteria:

* at risk for seizures or suspected to be having seizures;
* all seizure aetiologies except correctable metabolic abnormalities such as hypoglycaemia and hypocalcaemia;
* Term neonates (corrected gestational age between 35 and 44 weeks, postnatal age less than 28 days);
* weight > 2200g.
* Parental ability to comprehend and provide written informed consent

Exclusion Criteria:

* Cumulative seizure burden of 8 minutes/ hour or more in phases 1 and 2, Cumulative seizure burden of 30 minutes/hour or more in phase 3;
* Renal failure defined as anuria in the first 24 hours of life;
* Subjects in whom death seems imminent;
* Seizures caused by correctable metabolic abnormality, such as hypocalcaemia, hypoglycaemia.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the maximum safe and tolerated dose of Levetiracetam | 4 years
  A continual reassessment method will be used to determine the maximal safe and tolerated dose

SECONDARY OUTCOMES:
Levetiracetam CL | 4 years
  Population pharmacokinetic parameters for LEV Clearance (CL)will be calculated
Levetiracetam Vd | 4 years
  Population pharmacokinetic parameters for LEV Volume of distribution (Vd) will be calculated
Adverse event rates | 4 years
  Rates of adverse events seen with high dose LEV treatment will be reported and compared to rates seen in PHB control arm.
Long-term outcome | 8 years
  Rates of adverse long-term outcome ( Death or Disability at 24 months) will be compared between treatment arms
Seizure burden reduction | 4 years
  Number of patients with at least 50% seizure burden reduction post treatment will be compared between randomized treatment arms
Seizure freedom rates | 4 years
  Number of patients who become seizure free for 24 hours post treatment will be compared between the randomized treatment groups in each stage of the study
Estimate of efficacy of higher dose LEV | 4 years
  Assuming no dose limiting toxicity is demonstrated and the study proceeds to completion, 50 subjects will be treated at 120mg/kg or higher dosing level. This sample size will give satisfactory power for estimating additional efficacy of higher doses. For example, if we document an additional response rate of 15%, this sample size will provide a 95% confidence interval (0.051, 0.248) around that estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Sonya G Wang, M.D., Principal Investigator — University of Minnesota; Cynthia M Sharpe, M.D., Principal Investigator — Auckland City Hospital; Jeff J Gold, M.D. PhD, Principal Investigator — University of California, San Diego; Richard H Haas, MBBChir, Principal Investigator — University of California, San Diego
Locations (5):
- United States (2):
  - University of California, San Diego, San Diego, California
  - University of Minnesota, Minneapolis, Minnesota
- New Zealand (3):
  - Auckland City Hospital, Auckland, Auckland
  - Middlemore Hospital, Auckland, Auckland
  - Capital and Coast District Health Board, Te Whatu Ora, Health New Zealand, Wellington, Wellington Region

IPD SHARING:
Plan to Share IPD: No